CLINICAL TRIAL: NCT05204147
Title: A Phase I Study of Actinium-225 Labeled Humanized Anti-CEA M5A Antibody in Patients With CEA Producing Advanced or Metastatic Cancers
Brief Title: Actinium 225 Labeled Anti-CEA Antibody (Ac225-DOTA-M5A) for the Treatment of CEA Producing Advanced or Metastatic Cancers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20449; NCI-2021-14101 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20449 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH)
Record Dates: First submitted 2022-01-11; First posted 2022-01-24 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-03

CONDITIONS: Advanced Cancer; Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Ac225-DOTA-M5A) (Experimental): Patients receive Ac225-DOTA-M5A IV over 25 minutes on day 1.
  Interventions: Drug: Actinium Ac 225-DOTA-anti-CEA Monoclonal Antibody M5A; Procedure: Biospecimen Collection

INTERVENTIONS:
Drug: Actinium Ac 225-DOTA-anti-CEA Monoclonal Antibody M5A — Given IV
  Other Names: 225Ac-DOTA-anti-CEA Monoclonal Antibody M5A; 225Ac-DOTA-M5A Humanized Anti-CEA Antibody
Procedure: Biospecimen Collection — Correlative studies
  Other Names: Biological Sample Collection; Biospecimen Collected

SUMMARY:
This phase I study tests the safety, side effects, and best dose of Ac225-DOTA-M5A in treating patients with CEA positive colorectal cancer that has spread to other places in the body (advanced). Ac225-DOTA-M5A is a humanized monoclonal anti-CEA antibody, linked to a radioactive agent called actinium 225. M5A attaches to CEA positive cancer cells in a targeted way and delivers actinium 225 to kill them.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To establish the maximum tolerated dose (MTD) of actinium Ac 225-DOTA-anti-CEA Monoclonal Antibody M5A (225Ac-DOTA-M5A) humanized anti-carcinoembryonic antigen (CEA) antibody when given intravenously and to describe the toxicities at each dose studied.

SECONDARY OBJECTIVES:

I. To begin to evaluate the clinical activity of the agent in metastatic colorectal cancer.

II. To evaluate the organ biodistribution, pharmacokinetics and organ dose estimates of 225Ac-DOTA-M5A.

OUTLINE: This is a dose-escalation study.

Patients receive Ac225-DOTA-M5A intravenously (IV) over 25 minutes on day 1.

After completion of study treatment, patients are followed weekly for 6-10 weeks, and then medical records are reviewed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologic diagnosis of a malignancy that expresses CEA. If biopsies were performed at an outside facility, the histology must be reviewed and confirmed by the Department of Pathology at the City of Hope
* Patients must have tumors that produce CEA as documented by either an elevated serum CEA above the institutional limit of normal or by immunohistochemical methods. Positive CEA immunohistochemical staining, for the purposes of this protocol, is graded 0-3 and the percentage of tumor cells positive is estimated. A positive CEA stain is determined if more than 30% of the tumor cells have an intensity of 2+ or greater
* Patients must have an advanced disease for which no standard or effective treatment is available. Patients who refuse a standard but non-curative treatment is available may also be considered
* Karnofsky performance status >= 60% and an estimated survival of at least 3 months
* Patients must be >= 18 years old as phase I data for the antibody is not available for younger patients.
* The effects of Ac-225-DOTA-M5A on the developing fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation. Should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* Adequate bone marrow function as evidenced by white blood count (WBC) >= 4000/ul, absolute neutrophil count >= 1500/ul, platelet count >= 125,000/ul are required
* Adequate renal function as evidenced by a creatinine =< 1.5 mg/dl and/or a calculated creatinine clearance >= 60 cc/min
* Adequate liver function as evidenced by bilirubin =< 1.5 mg/dl and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) no greater than 2 times the upper limit of normal. Less than 1/3 of the liver must be estimated to be involved with tumor
* Presence of measurable disease is required for study entry
* All patients must be seen in consultation by City of Hope Radiation Oncology and City of Hope Medical Oncology prior to entry onto this trial
* All subjects must have the ability to understand and the willingness to sign a written informed consent
* Prior radiotherapy, immunotherapy, or chemotherapy must have been completed at least 4 weeks prior to patient entry on this study (6 weeks if treated with mitomycin-c or nitrosoureas) and patients must have recovered from any expected side effects of prior therapy

Exclusion Criteria:

* Patients should not have any uncontrolled illness including ongoing or uncontrolled active infection
* Patients may not be receiving any other investigational agents, or concurrent biological, chemotherapy, or radiation therapy
* Pregnant women are excluded from this study because Ac225-DOTA-M5A are agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Ac225-DOTA-M5A, breastfeeding should be discontinued if the mother is treated with Ac225-DOTA-M5A
* Patients with recurrent or progressive brain or leptomeningeal involvement with cancer. Patients that have had previous therapies for brain metastasis or leptomeningeal disease with demonstrated response or stable disease at least four weeks after therapy will be eligible for the trial
* Patients who have received previous radiation to > 50% of their bone marrow
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-06-02 (Actual); Primary Completion 2026-07-21 (Estimated); Study Completion 2026-07-21 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 6 months
  The toxicities observed at each dose level will be summarized in terms of type (organ affected or laboratory determination such as absolute neutrophil count), severity (by National Cancer Institute Common Toxicity Criteria and nadir or maximum values for the laboratory measures), time of onset (i.e. course number), and attribution to study drug. Tables will be created to summarize these toxicities and side effects by dose and by course.
Maximum tolerated dose (MTD) | Up to 36 months
  The MTD is defined as the highest dose tested in which fewer than 33% of patients experienced dose limiting toxicities (DLT) attributable to the study drugs, when at least six patients were treated at that dose and are evaluable for toxicity. The MTD is one dose level below the DLT-level. At least 6 patients will be treated at the MTD.

SECONDARY OUTCOMES:
Overall survival | Assessed up to 6 months
  From first day of treatment to time of death due to any cause.
Progression-free survival | Assessed up to 6 months
  From first day of treatment to the first observation of disease progression or death due to any cause.
Time to failure | Assessed up to 6 months
  From first day of treatment to the first observation of disease progression or death due to disease.
Best overall response | Up to 6 months
  Evaluated with complete response, partial response, progressive disease or stable disease. The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The patient's best response assignment will depend on the achievement of measurement criteria, but confirmation is not necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Y Wong, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States